CLINICAL TRIAL: NCT01059019
Title: Epithelial Healing and Visual Outcomes of Patients Using Omega-3 Supplements as an Adjunct Therapy Before and After Photorefractive Keratectomy (PRK) Surgery
Brief Title: Epithelial Healing and Visual Outcomes Using Omega-3 Therapy Before and After Photorefractive Keratectomy (PRK) Surgery
Acronym: Omega-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, David J Schanzlin, DSchanzlin, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 091487
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Refractive Error
Keywords: Refractive Surgery; PRK; Photorefractive Keratectomy; Omega 3 Fatty Acids; Cornea
MeSH Terms: conditions — Refractive Errors; Corneal Diseases | interventions — Carboxymethylcellulose Sodium; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator): Twenty patients labeled as group A (Control Group) will not receive the omega-3 supplement. The Control Group will be treated in the same standard professional way as our normal refractive patients.
  Interventions: Dietary Supplement: Omega-3 Fatty Acid Supplements
- Treatment (Experimental): 20 patients labeled as group B (Treatment group) will be given omega- 3 supplements 1 capsule 3 x a day for 2 weeks pre op and 1 month post op plus the regular post op medications. From these supplements, this will be equivalent to 750 mg of omega 3 fatty acids (both EPH and DHA), 1000 mg of Flaxseed oil, and about 183 IU of vitamin E per day
  Interventions: Dietary Supplement: Omega-3 Fatty Acid Supplements

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acid Supplements — Twenty patients labeled as group A (Control Group) will not receive the omega-3 supplement. The Control Group will be treated in the same standard professional way as our normal refractive patients, while another 20 patients labeled as group B (Treatment group) will be given omega- 3 supplements 1 capsule 3 x a day for 2 weeks pre op and 1 month post op plus the regular post op medications. From these supplements, this will be equivalent to 750 mg of omega 3 fatty acids (both EPH and DHA), 1000 mg of Flaxseed oil, and about 183 IU of vitamin E per day. Patients will be asking to follow up postoperatively after 2 days, 4 days, 1 week, 3 months and 6 months
  Other Names: TheraTears; Omega 3

SUMMARY:
The purpose of this study is to demonstrate that omega-3 supplement can be use as an adjunct therapy for PRK patients. The investigators believe that omega-3 supplement will reduce the size of persistent epithelial defects (PEDS) and eventually hasten the corneal reepithelialization after PRK surgery. If the outcome of this study proves to be effective, then PRK would be a more attractive option to those seeking refractive treatment.

DETAILED DESCRIPTION:
Dry eye and persistent epithelial defects (PEDS) following LASIK and PRK are one of the most common conditions encountered by refractive surgeons and their patient's today.¹-⁴ They are associated with significant clinical morbidity in patients resulting in minor problems such as discomfort, to extreme debilitation such as visual loss. There is no accepted definition of persistent epithelial defect (PED) that includes a time period of recovery. We favor the definition given in one text "… when the epithelium fails to re-grow over a defect within the expected time course.⁵ The causes of PED are diverse, with several definite etiologies' including dry eyes, limbal stem cell deficiency, diabetes mellitus and neurotrophic problems. A variety of treatment modalities have been described for PED. The elimination of predisposing associated risk remains a key factor in the management process. Therefore, to prevent and manage this common disorder it is important to have an understanding of the pathophysiology of dry eye after LASIK and PRK. This includes and understanding of the relationship and interaction between inflammation, sensory denervation and essential fatty acid pathways. Reports of clinical efficacy of anti-inflammatory therapies for treatment of dry eye disease provide direct proof of the principle that inflammation is involved in the etiology of dry eye disease. Research has shown that the omega-3 polyunsaturated fatty acids are some of the most effective natural anti inflammatory agents available. The active ingredients in omega 3, EPA ( Eicosapentanoic acid ) which is a 20 carbon omega 3-fatty acid with 5 double-bonds , and DHA ( docosahexanoic acid )which is 22 carbon omega-3 fatty acid with 6 double bond, both found in certain fish oils enhance the conversion of COX ( cyclooxygenase) to prostaglandin E3. A natural anti inflammatory agent, prostaglandin E3 competitively inhibits the effects of the arachidonic acid conversion to prostaglandin E2, a highly inflammatory substance. Prostaglandin E3 also inhibits the synthesis of TNFα and IL-1β, both of which are inflammatory leukotrienes, also by competitive inhibition.⁶ʹ⁷ By decreasing inflammation and stimulating aqueous tear production in rabbits cAMP has been shown to stimulate aqueous tear secretion in dry eye. Furthermore, by decreasing inflammation and augmenting oil and water layers of the tear film, omega-3 supplementation with fish oil rich in EPA may improve both the lipid and aqueous component of the tear film. This may improve surgical outcomes by stabilizing the tear film, reducing epithelial defects and promoting wound healing

ELIGIBILITY:
Inclusion Criteria:

* Male or female candidate for PRK with refractive error of -1.00 to -6.00
* Male or female 18- 28 (may consider increasing this range) years old and >60 years old post cataract surgery for enhancement.
* Patients without history of diabetes.
* Patients without history of hemorrhagic stroke.
* Patient without history of blood dyscrasia.
* Patient without history of diarrhea, abdominal bloating, and indigestion.
* Patient without history of peptic ulcer disease, gastroesophageal reflux and gastroesophageal reflux disease.

Exclusion Criteria:

* Male or female < 18 years old for PRK.
* Male or female with a refractive error < -1.00 or >-6.00
* Patient with history of diabetes.
* Patient with history of hemorrhagic stroke.
* Patient with history of Blood dyscrasia.
* Patient with history of peptic ulcer disease, gastroesophageal reflux and gastroesophageal reflux disease.
* Patient with history of diarrhea, abdominal bloating and indigestion.
* Pregnant women and women that are lactating (nursing mothers)

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Visual acuity, tear break up time, and corneal uptake will be assessed. Photographs will be taken. Calculation of the area in diameter will be assessed using Adobe Photoshop. Comparisons between each group will be made. | 2 and 4 days, 1 week, 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: David J Schanzlin, MD, Principal Investigator — UCSD Shiley Eye Center
Locations (1):
- UCSD Shiley Eye Center, La Jolla, California, United States

REFERENCES:
- [Background] Kanellopoulos AJ, Pallikaris IG, Donnenfeld ED, Detorakis S, Koufala K, Perry HD. Comparison of corneal sensation following photorefractive keratectomy and laser in situ keratomileusis. J Cataract Refract Surg. 1997 Jan-Feb;23(1):34-8. doi: 10.1016/s0886-3350(97)80148-4. PMID 9100105
- [Background] Linna TU, Vesaluoma MH, Perez-Santonja JJ, Petroll WM, Alio JL, Tervo TM. Effect of myopic LASIK on corneal sensitivity and morphology of subbasal nerves. Invest Ophthalmol Vis Sci. 2000 Feb;41(2):393-7. PMID 10670467
- [Background] Chuck RS, Quiros PA, Perez AC, McDonnell PJ. Corneal sensation after laser in situ keratomileusis. J Cataract Refract Surg. 2000 Mar;26(3):337-9. doi: 10.1016/s0886-3350(99)00416-2. PMID 10713225
- [Background] Albietz JM, Lenton LM, McLennan SG. Effect of laser in situ keratomileusis for hyperopia on tear film and ocular surface. J Refract Surg. 2002 Mar-Apr;18(2):113-23. doi: 10.3928/1081-597X-20020301-02. PMID 11934197
- [Background] Poon AC, Geerling G, Dart JK, Fraenkel GE, Daniels JT. Autologous serum eyedrops for dry eyes and epithelial defects: clinical and in vitro toxicity studies. Br J Ophthalmol. 2001 Oct;85(10):1188-97. doi: 10.1136/bjo.85.10.1188. PMID 11567963
- [Background] Maroon JC, Bost JW, Borden MK, Lorenz KM, Ross NA. Natural antiinflammatory agents for pain relief in athletes. Neurosurg Focus. 2006 Oct 15;21(4):E11. doi: 10.3171/foc.2006.21.4.12. PMID 17112189
- [Background] Afonso AA, Sobrin L, Monroy DC, Selzer M, Lokeshwar B, Pflugfelder SC. Tear fluid gelatinase B activity correlates with IL-1alpha concentration and fluorescein clearance in ocular rosacea. Invest Ophthalmol Vis Sci. 1999 Oct;40(11):2506-12. PMID 10509643
- [Background] Prabhasawat P, Tseng SC. Frequent association of delayed tear clearance in ocular irritation. Br J Ophthalmol. 1998 Jun;82(6):666-75. doi: 10.1136/bjo.82.6.666. PMID 9797670
- [Background] Macsai MS. The role of omega-3 dietary supplementation in blepharitis and meibomian gland dysfunction (an AOS thesis). Trans Am Ophthalmol Soc. 2008;106:336-56. PMID 19277245
- [Background] Kotani N, Hashimoto H, Kushikata T, Yoshida H, Muraoka M, Takahashi S, Matsuki A. Intraoperative prostaglandin E1 improves antimicrobial and inflammatory responses in alveolar immune cells. Crit Care Med. 2001 Oct;29(10):1943-9. doi: 10.1097/00003246-200110000-00016. PMID 11588457
- [Background] Narumiya S, Sugimoto Y, Ushikubi F. Prostanoid receptors: structures, properties, and functions. Physiol Rev. 1999 Oct;79(4):1193-226. doi: 10.1152/physrev.1999.79.4.1193. PMID 10508233
- [Background] Pholpramool C. Secretory effect of prostaglandins on the rabbit lacrimal gland in vivo. Prostaglandins Med. 1979 Sep;3(3):185-92. doi: 10.1016/0161-4630(79)90102-2. PMID 233220
- [Background] Gilbard JP, Rossi SR, Heyda KG, Dartt DA. Stimulation of tear secretion by topical agents that increase cyclic nucleotide levels. Invest Ophthalmol Vis Sci. 1990 Jul;31(7):1381-8. PMID 2365569
- [Background] Ambrosio R Jr, Wilson SE. Complications of laser in situ keratomileusis: etiology, prevention, and treatment. J Refract Surg. 2001 May-Jun;17(3):350-79. doi: 10.3928/1081-597X-20010501-09. PMID 11383767
- [Background] Saad HA, Terry MA, Shamie N, Chen ES, Friend DF, Holiman JD, Stoeger C. An easy and inexpensive method for quantitative analysis of endothelial damage by using vital dye staining and Adobe Photoshop software. Cornea. 2008 Aug;27(7):818-24. doi: 10.1097/ICO.0b013e3181705ca2. PMID 18650669